CLINICAL TRIAL: NCT01346254
Title: Glucose Control in Pre-Diabetic Renal Transplant Patients: Efficacy and Safety of Vildagliptin and Pioglitazone
Brief Title: Glucose Control in Pre-Diabetic Renal Transplant Patients
Acronym: GCPD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Marcus Saemann (Other)
Responsible Party: Sponsor-Investigator, Marcus Saemann, Dr, Medical University of Vienna
Organization: Medical University of Vienna (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GCPD
Record Dates: First submitted 2011-04-29; First posted 2011-05-02 (Estimated); Last update posted 2011-12-05 (Estimated); Status verified 2011-12

CONDITIONS: Impaired Glucose Tolerance; Kidney Transplantation
Keywords: after
MeSH Terms: conditions — Glucose Intolerance | interventions — Vildagliptin; Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Vildagliptin (Experimental): 16 patients randomized into this arm will receive vildagliptin (Galvus) 50mg orally once daily
  Interventions: Drug: Vildagliptin; Behavioral: Life-Style Modification
- Pioglitazone (Experimental): 16 patients randomized into this arm will receive pioglitazone (Actos) 30mg orally once daily
  Interventions: Drug: Pioglitazone; Behavioral: Life-Style Modification
- Placebo (Placebo Comparator): 16 patients randomized into this arm will receive placebo medication orally once daily
  Interventions: Behavioral: Life-Style Modification

INTERVENTIONS:
Drug: Vildagliptin — 50mg tablets once daily 20 min before breakfast for 3 months
  Other Names: Galvus
  Arms: Vildagliptin
Drug: Pioglitazone — 30mg tablets once daily 20 min before breakfast for 3 months
  Other Names: Actos
  Arms: Pioglitazone
Behavioral: Life-Style Modification — All study participants were counselled regarding life-style modification including regular exercise, weight loss and diet.

SUMMARY:
Development of New-Onset Diabetes after Transplantation (NODAT) is common and serious complication after kidney transplantation. Patients who develop NODAT are at increased risk for loss of the transplanted organ and for diseases of the cardiovascular system.

It is believed that in many patients the development of overt NODAT is preceded by a phase of impaired glucose tolerance that is called pre-diabetes.

This study aims at improving glucose metabolism in patients after kidney transplantation who are in a pre-diabetic metabolic state. Patients who exhibit impaired glucose tolerance (IGT) after kidney transplantation are randomized to either receive vildagliptin (Galvus), pioglitazone(Actos) or placebo for three months.

The investigators hypothesize that treatment with vildagliptin or pioglitazone leads to improved glycemic control compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Time since renal transplantation > 6 months
* Stable graft function
* Routine OGTT has been performed, and pre-diabetes has been diagnosed by pathological OGTT (2h, 75 g glucose, glucose level between 140 and 200 mg/dl)
* Informed consent of the patient

Exclusion Criteria:

* Patients with type 1 or type 2 diabetes
* Patients with NODAT (2h glucose level at OGTT >200 mg/dl)
* allergy against vildagliptin or pioglitazone
* pregnancy
* GFR<15ml/min/1.73 with need for dialysis
* hepatic impairment

Ages: 18 Years to 81 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2009-12; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Oral glucose tolerance test (OGTT) | three months
  Glucose tolerance and insulin resistance three months after study start will be measured by means of a frequent sampling OGTT (75g glucose, determination of glucose, insulin and C-peptide) over 120 mins.

SECONDARY OUTCOMES:
glycated hemoglobin | 3 months
  HbA1c will be measured after three months and compared between the study arms
Renal function | 3 months
  Renal function will be assessed by measuring serum creatinin and glomerular filtration rate (GFR)at the beginning of the study and after three months of treatment
Liver function | 3 months
  Liver enzymes (ALAT, ASAT, Gamm-GT) will be measured at the start of the study and after three months treatment
Lipid profiles | 3 months
  Lipid profiles will be analyzed at the beginning and end of the study including Cholesterol, HDL, LDL and triglycerides.

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Säemann, MD, Principal Investigator — Medical University of Vienna, Department of Internal Medicine III, Division of Nephrology and Dialysis
Locations (1):
- Allgemeines Krankenhaus der Stadt Wien, Universitätskliniken, Vienna, Austria

REFERENCES:
- [Derived] Lo C, Toyama T, Oshima M, Jun M, Chin KL, Hawley CM, Zoungas S. Glucose-lowering agents for treating pre-existing and new-onset diabetes in kidney transplant recipients. Cochrane Database Syst Rev. 2020 Jul 30;8(8):CD009966. doi: 10.1002/14651858.CD009966.pub3. PMID 32803882